CLINICAL TRIAL: NCT05770401
Title: Internet-Behavioral Cough Suppression Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Montana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 163-22
Record Dates: First submitted 2023-02-01; First posted 2023-03-15 (Actual); Results first posted 2025-06-05 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2024-01

CONDITIONS: Cough; Chronic Disease
Keywords: refractory chronic cough; behavioral cough suppression therapy
MeSH Terms: conditions — Cough; Chronic Disease; Chronic Cough

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internet-Behavioral Cough Suppression Therapy (Experimental): Participants will watch treatment-specific educational and training videos and perform the training exercises as recommended. There are a total of five videos ranging from 2-5 minutes in length. Participants will be asked to watch the videos at least once weekly. Daily training exercises will be discussed in the videos and should take no more than a few minutes to complete every day. All exercises are non-invasive and are not physically demanding. Each week participants will complete a progress check question that will take less than one minute to answer, indicating whether they are watching the videos and completing the exercises as recommended.
  Interventions: Behavioral: Internet-Behavioral Cough Suppression Therapy
- Sham Treatment (Sham Comparator): Participants will watch sham treatment-specific educational and training videos and perform the training exercises as recommended. There are a total of five videos ranging from 2-5 minutes in length. Participants will be asked to watch the videos at least once weekly. Daily training exercises will be discussed in the videos and should take no more than a few minutes to complete every day. All exercises are non-invasive and are not physically demanding. Each week participants will complete a progress check question that will take less than one minute to answer, indicating whether they are watching the videos and completing the exercises as recommended.
  Interventions: Behavioral: Sham Treatment

INTERVENTIONS:
Behavioral: Internet-Behavioral Cough Suppression Therapy — Participants will access training modules to learn behavioral techniques and will implement them in daily life over a four-week period.
  Arms: Internet-Behavioral Cough Suppression Therapy
Behavioral: Sham Treatment — Participants will access training modules to learn behavioral techniques and will implement them in daily life over a four-week period.
  Arms: Sham Treatment

SUMMARY:
The goal of this randomized, placebo-controlled, clinical trial is to develop and test the efficacy of an Internet-based behavioral intervention for refractory chronic cough. The main questions it aims to answer are:

* What are the best recruitment pathways to find people living with refractory chronic cough in Montana?
* Is Internet-Behavioral Cough Suppression Therapy (iBCST) efficacious?
* Do iBCST participants find it satisfactory?
* Is using Hyfe research app to monitor cough frequency feasible in rural areas?

Participants will complete iBCST or a placebo treatment virtually. Some participants will take part in qualitative interviews and use Hyfe research app for ambulatory cough frequency monitoring.

ELIGIBILITY:
Inclusion Criteria:

* No barriers to using a computer or smartphone (e.g., no significant fine motor or visual problems).
* Internet and e-mail access and the ability to use it.
* Suffering from a cough lasting at least eight weeks that is:
* Largely unproductive (cough up no more than a few teaspoons worth of clear or white sputum or mucus in a 24-hour period).
* Report of cough triggered by identifiable stimuli including and not limited to any combination of the following: cold air, talking, laughing, taking a deep breath, exercise, crumbly foods, strong smells or odors, fumes from paint or cleaning sprays.
* Often preceded by the sensation of an urge-to-cough (e.g., tickle or itch) at the level of the throat.
* Self-report of receiving the following assessments for current cough symptoms with unremarkable results:
* Physical evaluation by at least one physician.
* Chest x-ray.
* Willingness to avoid other potential cough treatments during the course of the study (or alert study personnel if alternative treatment is implemented out of necessity).

Exclusion Criteria:

* Current smoker of any substance.
* Diagnosis of any of the following:
* Respiratory disease (e.g., chronic obstructive pulmonary disease, asthma)
* Neurogenic disease (e.g., Parkinson's disease, cerebrovascular disease)
* Head and neck cancer
* Self-report of difficulty swallowing since having chronic cough
* Use of the following medication:
* Angiotensin-converting enzyme inhibitor (ACE-I) in the past four weeks: benzapril (Lotensin), Captopril (Capoten), Enalapril/Enalaprilat (Vasotec oral and injectable), Fosinopril (Monopril), Lisinopril (Zestril and Prinivil), Moexipril (Univasc), Perindopril (Aceon), Quinapril (Accupril), Ramipril (Altace), and Trandolapril (Mavik).
* Use of a neuromodulator medication in the past 48 hours: Neurontin (Gabapentin) and amitriptyline.
* Individuals with dysphonia (abnormal voice; either self-reported or perceived by study personnel during enrollment interview) will be excluded unless they have had a normal laryngoscopy (endoscopic assessment of the larynx) by an otolaryngologist (ENT) within the past year specifically for their cough.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jane Reynolds, PhD, Principal Investigator — Assistant Professor
Locations (1):
- University of Montana, Missoula, Montana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Individuals with refractory chronic cough in the United States were recruited for the study via social media campaigns, newspaper advertisements, flyers sent to voice and upper airway clinics, word-of-mouth, and Facebook support groups. Recruitment took place from May 2023-2024.
Period: Overall Study
Arm/Group | Internet-Behavioral Cough Suppression Therapy | Sham Treatment
Started | 23 | 16
Completed | 18 | 12
Not Completed | 5 | 4
Not completed — Lost to Follow-up | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Internet-Behavioral Cough Suppression Therapy | Sham Treatment | Total
Number analyzed (Participants) | 23 | 16 | 39
Age, Continuous [Mean (Standard Deviation); unit: Age] — Population: Five IBCST participants and four control participants did not complete the intervention and no post-treatment data was collected from them so they are not included in any analyses.
  Age | 61.2 (9.4) | 59.3 (8.5) | 60.5 (9)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Five IBCST participants and four control participants did not complete the intervention and no post-treatment data was collected from them so they are not included in any analyses.
  Participants
    Female | 21 | 13 | 34
    Male | 2 | 3 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Five IBCST participants and four control participants did not complete the intervention and no post-treatment data was collected from them so they are not included in any analyses.
  Participants
    Hispanic or Latino | 0 | 0 | 0
    Not Hispanic or Latino | 23 | 16 | 39
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Five IBCST participants and four control participants did not complete the intervention and no post-treatment data was collected from them so they are not included in any analyses.
  Participants
    American Indian or Alaska Native | 0 | 1 | 1
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 0 | 1 | 1
    White | 23 | 14 | 37
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Leicester Cough Questionnaire
Description: Cough-related quality of life will be measured with the Leicester Cough Questionnaire (LCQ), a valid, reliable, and repeatable measure of cough-related quality of life. The LCQ is a 19-item questionnaire containing physical, psychological, and social domains. Scores for the LCQ include mean scores for each domain (ranging from 1 to 7) and a total score calculated as the sum of the domain scores (ranging from 3 to 21). A higher score indicates better quality of life. A change in 1.3 is considered clinically significant. The LCQ total score was the primary outcome measure in this study.
Time Frame: Pre-treatment, one-week post-treatment, one-month post-treatment
Population: One participant in the IBCST group was lost to follow up at one-month post-treatment and values are missing.
Measure: Mean (Standard Deviation); unit: Total LCQ Score
Arm/Group | Internet-Behavioral Cough Suppression Therapy | Sham Treatment
Number analyzed (Participants) | 18 | 12
Total LCQ Score
  Pre-intervention | 9.04 (7.32) | 8.86 (7.6)
  One-week post-treatment | 12.78 (12.89) | 9.44 (12.27)
  one-month post-treatment: number analyzed (Participants) | 17 | 12
  one-month post-treatment | 13.04 (4.31) | 9.70 (18.38)
Statistical Analysis 1: Comparison: Internet-Behavioral Cough Suppression Therapy vs Sham Treatment; The null hypothesis was there would be no significant difference in LCQ total score change from baseline to one-week post-treatment between groups; Test type: Superiority; p = .014, ANCOVA; Mean Difference (Final Values) = 3.24, 95% CI 2-sided [.72 to 5.76], Standard Error of Mean 1.227

2. Secondary Outcome: Cough Severity Visual Analog Scale
Description: Cough Severity Visual Analog Scale (VAS) is a 100-millimeter line with anchors of 0 "no problem" and 100 "worst possible problem" where participants place a mark to represent the severity of their current cough problem. A reduction of at least 30-millimeters is considered clinically meaningful for the Cough Severity VAS.
Time Frame: Pre-intervention, one-week post-treatment, one-month post-treatment
Population: One participant in the IBCST group was lost to follow up at one-month post-treatment and values are missing.
Measure: Mean (Standard Deviation); unit: VAS Total Score
Arm/Group | Internet-Behavioral Cough Suppression Therapy | Sham Treatment
Number analyzed (Participants) | 18 | 12
VAS Total Score
  Pre-intervention | 49 (15.97) | 49.08 (22.39)
  One-week post-treatment | 33.94 (21.32) | 50.08 (22.39)
  One-month post-treatment: number analyzed (Participants) | 17 | 12
  One-month post-treatment | 44.18 (22.85) | 56.42 (23.74)
Statistical Analysis 1: Comparison: Internet-Behavioral Cough Suppression Therapy vs Sham Treatment; The null hypothesis was there would be no significant difference in Cough Severity VAS Scores from baseline to one-week post-treatment between groups; Test type: Superiority; p = .056, ANCOVA; Mean Difference (Final Values) = -16.1, 95% CI 2-sided [-32.7 to 0.46], Standard Error of Mean 8.804

ADVERSE EVENTS:
Time Frame: From enrollment to one-month post-treatment.
Description: This was a behavioral intervention with essentially no risks to participants.
Arm/Group | Internet-Behavioral Cough Suppression Therapy | Sham Treatment
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/16
Other Adverse Events (participants affected / at risk) | 0/23 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-04-07): https://cdn.clinicaltrials.gov/large-docs/01/NCT05770401/Prot_SAP_000.pdf